CLINICAL TRIAL: NCT03583307
Title: Efficacy and Safety of Sirolimus in the Treatment of the Complicated Vascular Anomalies
Brief Title: Efficacy and Safety of Sirolimus to Vascular Anomalies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-618
Record Dates: First submitted 2018-06-17; First posted 2018-07-11 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Vascular Anomaly
Keywords: Sirolimus; Vascular anomalies
MeSH Terms: conditions — Vascular Malformations | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus was initiated at a dosage of 0.8 mg/m2 administered twice daily. Subsequently, the sirolimus dosage was adjusted monthly to achieve trough levels between 10 and 15 ng/mL.
  Other Names: Rapamycin

SUMMARY:
To evaluate the safety and efficacy of Sirolimus in complicated vascular anomalies in Chinese children

DETAILED DESCRIPTION:
Vascular anomalies are composed of vascular tumors and vascular malformations. The prognosis of vascular anomalies is significantly variable. Most of them had a benign course. However, complicated vascular anomalies can lead to disfigurement, organ disfunction and life-threatening with significant morbidity and mortality. Traditional treatments, including steroids, vincristine, cyclophosphamide and surgery, had limited response to complicated vascular anomalies. In the past few years, the inhibitor of the mammalian target of rapamycin (mTOR) signaling pathway-sirolimus has emerged as a treatment for severe vascular anomalies. Besides, preclinical studies also showed that the Phosphoinositide 3-kinase (PI3K)/protein kinase B (Akt)/mTOR pathway play an important role in the development of vascular tumors and vascular malformations. However, the exact efficacious rate and complications of sirolimus are still unknow in china because of the lack of large scale of prospective studies. Therefore, it's important to perform this prospective study to determine the safety and efficacy of sirolimus in the treatment of Chinese children with complicated vascular anomalies, and this study will also make contributions to the diagnoses and treatments of vascular anomalies.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the present research must be diagnosed with one of the following vascular anomalies:

  1. Kaposiform Hemangioendotheliomas without Kasabach-Merritt Phenomenon
  2. Tufted Angioma without Kasabach-Merritt Phenomenon
  3. Capillary Malformations
  4. Lymphatic Malformations
  5. Venous Malformations
  6. Capillary-Venous Malformation (CVM)
  7. Capillary-Lymphatic Malformation (CLM)
  8. Lymphatic-Venous Malformation (LVM)
  9. Capillary-Lymphatic-Venous Malformation (CLVM)
  10. Multifocal Lymphangiomatosis and Thrombocytopenia (MLT)
* Patients must be 0 - 18 years of age at the time of study entry.
* Without functional impairment requiring treatment of corticosteroid.
* Organ function requirements:
* Adequate liver function Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)for age, and alanine transaminase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 x upper limit normal (ULN) for age.
* Adequate renal function 0-5 years of age maximum serum creatinine (mg/dL) of 0.8 6-10 years of age maximum serum creatinine (mg/dL) of 1.0 11-15 years of age maximum serum creatinine (mg/dL) of 1.2 16-18 years of age maximum serum creatinine (mg/dL) of 1.5
* Adequate bone marrow function:

Absolute Neutrophil Count (ANC) greater than or equal to 1 x 10 to the ninth/Liter

* Consent of parents (or the person having parental authority in families): Signed and dated written informed consent.

Exclusion Criteria:

* Allergy to sirolimus or other rapamycin analogues.
* Allergy to sirolimus or other rapamycin analogues.
* Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of randomization.
* Patients must not be known to be Human Immunodeficiency Virus positive or known immunodeficiency. Testing is not required unless a condition is suspected.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
* Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of sirolimus.
* Patients who have a history of malignancy.
* Patients with an inability to participate or to follow the study treatment and assessment plan.
* Patients who have a history of treatment with sirolimus or other mTOR inhibitor.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Volumetric changes in complicated vascular anomalies to sirolimus | Baseline, 6, and 12 months
  Response to sirolimus treatment was measured by volumetric magnetic resonance imaging (MRI) analyses, which were performed at baseline and 6 and 12 months after treatment and were independently assessed by 2 radiologists. Changes in size of vascular anomalies were classified as further growth (increase of ≥10%), no change (<10% increase and <10% decrease), partial involution (decrease of ≥10% and <75%), nearly complete involution (decrease of ≥75% and <100%), or complete involution (100%).
  Photographs of the complicated vascular anomalies were taken at months 0, 3, 6 and 12 by a medical photographer.
  Complete/nearly complete resolution of the vascular anomalies at month 12 compared to baseline based on the intra-patient blinded centralized independent qualitative assessments of month 12 MRI.
The changes in the patient's symptoms and/or complications. | Baseline, 3, 6, and 12 months

SECONDARY OUTCOMES:
Quality of Life in patients by the Pediatric Quality of Life Inventory TM (PedsQLTM) 4.0 Generic Core Scales. | Baseline, 6, 12 months
  The PedsQL 4.0 Generic Core Scales encompass: 1) Physical Functioning (8 items), 2) Emotional Functioning (5 items), 3) Social Functioning (5 items), and 4) School Functioning (5 items), and were developed through focus groups and cognitive interviews. The PedsQL 4.0 Generic Core Scales are comprised of parallel child self-report (ages 5-18) and parent proxy-report formats (ages 0-18). A 5-point response scale is utilized across child self-report for ages 8 to 18 and parent proxy-report (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem). For patients between ages 5-7, the response scale is simplified to a 3-point scale (0=not at all a problem; 2=sometimes a problem; 4=a lot of a problem. Items are reverse-scored and linearly transformed to a 0 to 100 scale (0=100, 1=75, 2 =50, 3=25, 4=0). Scale Scores are computed as the sum of the items divided by the number of items answered.
Measuring the impact of vascular anomalies on family functioning by PedsQLTM 4.0 Family Impact Module (FIM). | Baseline, 6, 12 months
Frequency of adverse events as assessed by CTCAE v4.0 | Baseline, 3, 6, 12 months
Changes in plasma levels fibrinogen and/ or D-dimers | Baseline, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Chen S, Yang K, Zhou J, Zhang X, Jiang X, Xu X, Lu G, Qiu L, Kong F, Zhang Y. A prospective multicenter study of sirolimus for complicated vascular anomalies. J Vasc Surg. 2021 Nov;74(5):1673-1681.e3. doi: 10.1016/j.jvs.2021.04.071. Epub 2021 May 31. PMID 34082006